CLINICAL TRIAL: NCT00220285
Title: A Phase II Open-label Study of SH L 749 in Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphomas
Brief Title: Study for Evaluation of Efficacy and Safety of SH L 749 to Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Yakuhin Ltd.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91102; 305618
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Non-Hodgkin's Lymphoma; Lymphoma, B-Cell; Lymphoma, Low-Grade
Keywords: Antigen; CD20
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Zevalin (SH L 749 , BAY86-5128)
- Arm 2 (Experimental)
  Interventions: Drug: Zevalin (SH L 749 , BAY86-5128)

INTERVENTIONS:
Drug: Zevalin (SH L 749 , BAY86-5128) — 0,3mCi/kg
  Arms: Arm 1
Drug: Zevalin (SH L 749 , BAY86-5128) — 0,4mCi/kg
  Arms: Arm 2

SUMMARY:
The purpose of this study is to investigate the antitumor effect and safety of the product for relapsed or refractory indolent B-cell non-Hodgkin's lymphomas.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Platelet counts of >/= 100,000/mm3
* Absolute neutrophil counts of >/= 1,200/mm3
* Bone marrow involvement < 25%

Exclusion Criteria:

* Patients who received hematopoietic stem cell transplantation, including bone marrow transplantation, peripheral blood stem cell transplantation, etc.
* Patients presenting with marked bone marrow hypocellularity (any suspected bone marrow hypocellularity should be confirmed by bone marrow biopsy)
* Patients with previous myocardial infarction within the past 1 year, with heart disease that requires treatment or with pulmonary dysfunction
* Patients with serious concomitant diseases (cardiac failure, renal failure, etc.)

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-08; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Best overall response rates (the percentage of patients who achieved PR or better response) | After 9 weeks or 13 weeks
The incidence of critical toxicity | During treatment period

SECONDARY OUTCOMES:
Safety evaluation | During treatment period
Complete response (CR or CRu) rates | After 9 weeks or 13 weeks
Progression-free survival (PFS) | After end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Japan (9):
  - Nagoya, Aichi-ken
  - Kashiwa-shi, Chiba
  - Maebashi, Gunma
  - Kanazawa, Ishikawa-ken
  - Isehara-shi, Kanagawa
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Chuo-ku, Tokyo
  - Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Tobinai K, Watanabe T, Ogura M, Morishima Y, Hotta T, Ishizawa K, Itoh K, Okamoto S, Taniwaki M, Tsukamoto N, Okumura H, Terauchi T, Nawano S, Matsusako M, Matsuno Y, Nakamura S, Mori S, Ohashi Y, Hayashi M, Endo K. Japanese phase II study of 90Y-ibritumomab tiuxetan in patients with relapsed or refractory indolent B-cell lymphoma. Cancer Sci. 2009 Jan;100(1):158-64. doi: 10.1111/j.1349-7006.2008.00999.x. Epub 2008 Oct 24. PMID 19018755